CLINICAL TRIAL: NCT03013582
Title: A Prospective Randomized Trial Comparing Tendon Wrapping With Amniotic Membrane and Tenolysis Versus Tenolysis Alone for Treatment of Tendon Adhesions of the Hand and Wrist
Brief Title: Amniotic Membrane Wrapping and Tenolysis Versus Tenolysis Alone for Treatment of Tendon Adhesions of the Hand/Wrist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16D.538
Record Dates: First submitted 2016-12-20; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Tendinopathy; Adhesions Nos Postoperative; Scar; Fibrosis
MeSH Terms: conditions — Tendinopathy; Cicatrix; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Amnion wrapping + Tenolysis (Experimental): Standard surgical tenolysis + wrapping of the released tendon with amnion.
  Interventions: Biological: Amnion Tendon Wrapping; Procedure: Surgical Tenolysis
- Tenolysis control (Placebo Comparator): Standard surgical tenolysis alone
  Interventions: Procedure: Surgical Tenolysis

INTERVENTIONS:
Biological: Amnion Tendon Wrapping — Tendon is wrapped with the allograft
  Arms: Amnion wrapping + Tenolysis
Procedure: Surgical Tenolysis — Surgical release of peritendinous scarred tissue

SUMMARY:
Tendon adhesions of the hand remain a ubiquitous problem facing hand surgeons and hand therapists alike. Despite their commonality, no consensus exists as to the best means of preventing adhesions, or the most ideal methods to treat them once they have occurred. The purpose of this study is to compare patient outcomes after standard operative tenolysis performed for adhesions of the hand to outcomes after tenolysis with the use of allograft human amniotic membrane.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo operative tenolysis of the flexor and/or extensor tendons of the hand will be recruited. Our target enrollment is 40 patients (20 control plus 20 experimental), based on the power analysis detailed in the next paragraph. Enrolled patients will be randomized to either standard operative tenolysis, or tenolysis with placement of AlloWrap. Randomization will be performed by computerized random number generator. All surgeries will be performed by one senior fellowship-trained hand surgeon. Baseline measurements of total active motion (TAM), passive range of motion (PROM), and survey scores of the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) and Patient Rated Wrist Evaluation (PRWE) will be recorded pre-operatively. In addition, patients' pain level will be assessed using the visual analog scale (VAS) both at rest, and during the examination. These same values will be re-evaluated at post-operative follow-up visits at 2 weeks, 1 month, 3 months and 6 months. PROM will also be evaluated intra-operatively by the surgeon, and documented.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients deemed candidates for operative tenolysis of the hand or wrist
* Age ≥18

Exclusion Criteria:

* Patients younger than 18 years at the time of surgery;
* Any patient who would not be able or willing to comply with the protocol or perform assessments;
* Patients with medical conditions that may preclude placement of human biological membrane;
* Patients who have previously undergone tenolysis on the operative hand;
* Patients that will have multiple surgeries that are deemed as possible confounders, particularly those requiring an additional incision;
* Is physically or mentally compromised (i.e. being currently treated for a psychiatric disorder, senile dementia, Alzheimer's disease) in a manner that would compromise his or her ability to participate in the clinical study;
* Is a prisoner;
* Is a transient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Total Active Motion (TAM) | 6 months
Passive Range of Motion (PROM) | 6 months

SECONDARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) | 6 months
  Validated Outcome score/questionnaire specific to wrist function
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 6 months
  Validated Outcome score/questionnaire generalized to upper extremity conditions
Complications | 2 weeks, One month, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Culp, MD, Principal Investigator — Thomas Jefferson University-Philadelphia Hand Center; Michael P Gaspar, MD, Study Director — Thomas Jefferson University-Philadelphia Hand Center

REFERENCES:
- [Background] Vucekovich K, Gallardo G, Fiala K. Rehabilitation after flexor tendon repair, reconstruction, and tenolysis. Hand Clin. 2005 May;21(2):257-65. doi: 10.1016/j.hcl.2004.11.006. PMID 15882604
- [Background] Rouhani A, Tabrizi A, Ghavidel E. Effects of non-steroidal anti-inflammatory drugs on flexor tendon rehabilitation after repair. Arch Bone Jt Surg. 2013 Sep;1(1):28-30. Epub 2013 Sep 15. PMID 25207280
- [Background] Kohanzadeh S, Lugo L, Long JN. Safety of antiadhesion barriers in hand surgery. Ann Plast Surg. 2013 May;70(5):527-9. doi: 10.1097/SAP.0b013e31827eace2. PMID 23542850
- [Background] Fairbairn NG, Randolph MA, Redmond RW. The clinical applications of human amnion in plastic surgery. J Plast Reconstr Aesthet Surg. 2014 May;67(5):662-75. doi: 10.1016/j.bjps.2014.01.031. Epub 2014 Jan 31. PMID 24560801
- [Background] Wu YF, Tang JB. Apoptosis in adhesions and the adhesion-tendon gliding interface: relationship to adhesion-tendon gliding mechanics. J Hand Surg Am. 2013 Jun;38(6):1071-8. doi: 10.1016/j.jhsa.2013.03.012. Epub 2013 May 6. PMID 23660197
- [Background] Ozboluk S, Ozkan Y, Ozturk A, Gul N, Ozdemir RM, Yanik K. The effects of human amniotic membrane and periosteal autograft on tendon healing: experimental study in rabbits. J Hand Surg Eur Vol. 2010 May;35(4):262-8. doi: 10.1177/1753193409337961. Epub 2009 Aug 17. PMID 19687075
- [Background] Branford OA, Lee DA, Bader DL, Grobbelaar AO. The mechanics of flexor tendon adhesions. J Hand Surg Eur Vol. 2012 Jul;37(6):555-63. doi: 10.1177/1753193411432675. Epub 2011 Dec 14. PMID 22170243
- [Background] Gaspar MP, Abdelfattah HM, Welch IW, Vosbikian MM, Kane PM, Rekant MS. Recurrent cubital tunnel syndrome treated with revision neurolysis and amniotic membrane nerve wrapping. J Shoulder Elbow Surg. 2016 Dec;25(12):2057-2065. doi: 10.1016/j.jse.2016.09.013. Epub 2016 Oct 14. PMID 27751716